CLINICAL TRIAL: NCT02746107
Title: RCT Concerning the Intention to Prescribe/Take Oral Anticoagulants for Atrial Fibrillation Depending on the Number of Risk Diagrams (w Treatment +/- w/Out Treatment), and Number of Years (1 or 5) for the Estimation of the Risk of Stroke.
Brief Title: Intention to Prescribe/Take OAC Depending on the Number of Risk Diagrams , and Period for the Estimation of the Risk.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cristian Baicus (Other)
Responsible Party: Sponsor-Investigator, Cristian Baicus, Professor of Internal Medicine, Carol Davila University of Medicine and Pharmacy
Organization: Carol Davila University of Medicine and Pharmacy (Other)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: Studiul Cozia
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: shared decision making; oral anticoagulant; atrial fibrillation; stroke; decision to treat
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- risk presented on 1 diagram (Experimental): decision aid with risk of stroke presented on 1 diagram (risk under OAC treatment)
  Interventions: Other: decision aid
- risk presented on 2 diagrams (Active Comparator): decision aid with risk of stroke presented on 2 diagrams (one presenting risk without and one presenting risk with treatment)
  Interventions: Other: decision aid
- 1year risk estimate (Active Comparator): risk of stroke presented over a timeframe of 1 year
  Interventions: Other: decision aid
- 5year risk estimate (Experimental): risk of stroke presented over a timeframe of 5 years
  Interventions: Other: decision aid
- CHA2DS2-VASC risk score 1 (Other): CHA2DS2-VASC risk score =1
  Interventions: Other: decision aid
- CHA2DS2-VASC risk score 2 (Other): CHA2DS2-VASC risk score =2
  Interventions: Other: decision aid
- CHA2DS2-VASC risk score 3 (Other): CHA2DS2-VASC risk score =3
  Interventions: Other: decision aid
- CHA2DS2-VASC risk score 4 (Other): CHA2DS2-VASC risk score =4
  Interventions: Other: decision aid
- CHA2DS2-VASC risk score 5 (Other): CHA2DS2-VASC risk score =5
  Interventions: Other: decision aid
- prescription to virtual patient (Active Comparator): prescription is done for a virtual patient
  Interventions: Other: decision aid
- prescription to physician himself (Experimental): prescription is done to physician himself
  Interventions: Other: decision aid

INTERVENTIONS:
Other: decision aid — decision aid with one/two diagrams decision aid with risk over one/five years decision aid with CHA2DS2-VASC risk score 1 to 5 target of the prescription: patient / physician hinself

SUMMARY:
Randomized study concerning the effect of the number of risk diagrams (with treatment +/- without treatment), the period of stroke risk estimation (one year or five years) and the target of prescription (the patient with atrial fibrillation or the physician himself, imagining she/he has atrial fibrillation) on the intention to prescribe or not oral anticoagulation.

DETAILED DESCRIPTION:
Objectives:

To answer the questions:

1. Concerning the decision to prescribe (take) treatment on the basis of a decision aid, are there necessary both diagrams (that with risk without treatment, and that with risk under treatment), or it is enough only the second (risk under treatment, which normally gives all the needed information)?
2. Concerning the decision to prescribe (take) treatment, is it a difference between the effects of the presentation on decision aid of the risk of stroke for the next 1 year, and the presentation of the estimated risk of stroke for the next 5 years?
3. Is the decision different if physicians prescribe the anticoagulant treatment to patients, over if they should take it themselves?

Study: 2x3 factorial randomized controlled trial (RCT) for comparison:

1. Between the decision aid with 2 images (without treatment + with treatment) and the one with 1 image (risk only with treatment)
2. Between the effect of the presentation of the stroke risk chart for 1 year and the stroke risk chart for 5 years.
3. The decision to prescribe to patients over the decision to take the treatment themselves.

The comparison will be made for the spectrum of risks (scores CHA2DS2-VASC) from 1-5.

Sample size: was calculated a sample of 948 participants (474 + 474) for p = 0.05, power = 80% statistical difference between decisions of 5% (from 95% to 90%). The study does not have enough power neither to compare the 5 groups CHA2DS2-VASC (but we will make these comparisons with exploratory purpose), nor to test interactions.

Participants: physicians participating to the National Congress of Internal Medicine, physicians participating to courses, professional manifestations.

Randomization: randomization will be done on graph type (1 or 2 pictures), duration of risk estimate (1 year and 5 years) and the size of CHA2DS2-VASC risk score (1 to 5), and target prescription (patient or the doctor himself), a total of 40 possibilities. Randomization will be done in blocks of 40.

Participants will be asked to decide, depending on the risk chart, if the patient (or himself) will be treated, ignoring the risk of bleeding.

The chart will contain the pictogram according to the CHA2DS2-VASC risk score, without communicating the actual score, and the physician will have to make the decision to treat or not, depending on the perceived risk, and not on treatment guidelines.

No. questionnaire: first digit = number of risk diagrams (1 or 2); second digit = number of years for which the risk of stroke is calculated (1 or 5); third digit = CHA2DS2-VASC score (1-5). Ex: 253: 2 decision aid diagrams (with and without treatment), with an estimated risk of stroke for the next five years, in a patient with CHA2DS2-VASC score =3.

Effect (outcome): decision to treat / not to treat the patient / physician himself, with oral anticoagulants.

Statistical analysis: It will look for differences in bivariate analysis, and multivariate = logistic regression (dependent variable = treatment decision, the independent variables = number of charts, period for risk assessment (one or 5 years), prescription target (patient or the physician himself), CHA2DS2-VASC score, time from graduation, medical/teaching grade, working in hospital / ambulatory, the size of the city the physician works in, specialty, gender, age, if the physician has/had someone close with stroke (data from questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* physicians who prescribe anticoagulant treatment for atrial fibrillation (cardiology, internal medicine, family medicine, hematology) or who deal with patients with stroke (neurology, pathology) or bleeding (gastroenterology)

Exclusion Criteria:

* physicians who never prescribe anticoagulant treatments, or do not deal with patients with stroke or bleeding because of anticoagulants

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 968 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Baicus, PhD, Study Chair — Carol Davila University of Medicine and Pharmacy Bucharest - Colentina Hospital
Locations (1):
- Colentina Clinica Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Undecided
At the end, when published

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: all study participants were 968 (in all arms of this factorial RCT)
Period: Overall Study
Arm/Group | All Study Participants
Started | 968
2 Diagrams DA | 482
1 Diagram DA | 486
1year Risk Estimate | 483
5year Risk Estimate | 485
Target=Patient | 486
Target=Physician | 482
CHA2DS2-VASC Score = 1 | 195
CHA2DS2-VASC Score = 2 | 189
CHA2DS2-VASC Score = 3 | 195
CHA2DS2-VASC Score = 4 | 197
CHA2DS2-VASC Score = 5 | 192
Completed | 968
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: age: median (min, max): 39 (25, 83)
Groups:
- All Participants: all participants in the study (968)
Arm/Group | All Participants
Number analyzed (Participants) | 968
Age, Continuous [Median (Full Range); unit: years] | 39 [25 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 704
  Male | 264
Region of Enrollment [Number; unit: participants]
  Romania | 968

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Prescribed Oral Anticoagulants (OAC) According to the Number of Decision Aid Diagrams
Description: after regarding the risk diagram, the physician will decide to prescribe/take or not the treatment
Time Frame: after seeing the decision aid (5 min)
Measure: Number; unit: participants
Groups:
- One Diagram: decision aid with one diagram (risk under treatment)
  decision aid: decision aid with one/two diagrams
- Two Diagrams: classical decision aid with 2 diagrams (risk without treatment, and risk with treatment)
  decision aid: decision aid with one/two diagrams
Arm/Group | One Diagram | Two Diagrams
Number analyzed (Participants) | 486 | 482
participants | 400 | 406
Statistical Analysis 1: Comparison: One Diagram vs Two Diagrams; Test type: Non-Inferiority or Equivalence — details provided in the protocol. Noninferiority margin=+/-5%; p = 0.83, Chi-squared; Risk Difference (RD) = 0.5, 95% CI 2-sided [-4 to 5.4]

2. Other Pre Specified Outcome: Number of Participants Who Prescribed Oral Anticoagulants (OAC) According to the Timeframe for Risk Presentation (1 vs 5 Years)
Description: the proportion of physicians deciding to prescribe OAC after seeing risk estimation on 1 vs 5 years
Time Frame: 5 minutes
Measure: Number; unit: participants
Groups:
- 5 Years Risk Estimation on DA: participants had to prescribe or not OAC after seeing the risk estimated on 5 years
- 1 Year Risk Estimation on DA (CHA2D2S-VASC Score): participants deciding to prescribe or not OAC after seeing the stroke risk estimation on 1 year (classical CHA2D2S-VASC score)
Arm/Group | 5 Years Risk Estimation on DA | 1 Year Risk Estimation on DA (CHA2D2S-VASC Score)
Number analyzed (Participants) | 485 | 483
participants | 412 | 394
Statistical Analysis 1: Comparison: 5 Years Risk Estimation on DA vs 1 Year Risk Estimation on DA (CHA2D2S-VASC Score); details provided in protocol;; Test type: Superiority or Other; p = 0.187, Chi-squared; Risk Difference (RD) = 3.4, 95% CI 2-sided [-1.3 to 8.1] — (risk on 5y) - (risk on 1y)

3. Other Pre Specified Outcome: Number of Participants Who Prescribed Oral Anticoagulants (OAC) According to the Target of Prescription (Patient vs. Physician Himself)
Description: the participant physicians were randomized to prescribe to virtual patients or to imagine that the risk seen in the diagram was that of themselves
Time Frame: 5 min
Measure: Number; unit: participants
Groups:
- Prescription to Patient: the participant physician were randomized to prescribe OAC to virtual patients
- Prescription to Physician Himself: the participants had to imagine that they had atrial fibrillation, the risk from the diagram was theirs, and had to decide to take or not the OACs
Arm/Group | Prescription to Patient | Prescription to Physician Himself
Number analyzed (Participants) | 486 | 482
participants | 442 | 364
Statistical Analysis 1: Comparison: Prescription to Patient vs Prescription to Physician Himself; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Difference (RD) = 15.4, 95% CI 2-sided [10.8 to 20] — patient - (physicians themselves)
Statistical Analysis 2: Comparison: Prescription to Patient vs Prescription to Physician Himself; Test type: Superiority or Other; p < 0.001, Regression, Logistic; adjustment for age, gender, CHA2D2s-VASC score, nr of diagrams, nr of years, presence of someone close with stroke, graduation year, speciality; Odds Ratio (OR) = 3.28, 95% CI 2-sided [2.25 to 4.78]

4. Other Pre Specified Outcome: Number of Participants Who Prescribed Oral Anticoagulants (OAC) According to the CHA2D2s-VASC Risk Score
Description: The proportion of OAC prescription for the range 1-5 of CHA2D2s-VASC scores. CHA2D2S-VASC risk score ranges from 1-5, with higher scores indicating a greater risk of stroke.
Time Frame: 5 min
Measure: Number; unit: participants
Arm/Group | CHA2D2S-VASC Risk Score 1 | CHA2D2S-VASC Risk Score 2 | CHA2D2S-VASC Risk Score 3 | CHA2D2S-VASC Risk Score 4 | CHA2D2S-VASC Risk Score 5
Number analyzed (Participants) | 195 | 189 | 195 | 197 | 192
participants | 146 | 159 | 164 | 172 | 165
Statistical Analysis 1: Comparison: CHA2D2S-VASC Risk Score 1 vs CHA2D2S-VASC Risk Score 2; CHA2D2S-VASC risk score 1 was the reference; Test type: Superiority or Other; p = 0.034, Chi-squared; CHA2D2S-VASC risk score 1 was reference; Risk Difference (RD) = 9.3, 95% CI 2-sided [1.2 to 17] — positive value means higher proportion of prescription, CHA2D2S-VASC risk score 1 was reference
Statistical Analysis 2: Comparison: CHA2D2S-VASC Risk Score 1 vs CHA2D2S-VASC Risk Score 3; Test type: Superiority or Other; p = 0.033, Chi-squared; Risk Difference (RD) = 9.2, 95% CI 2-sided [1.2 to 17]
Statistical Analysis 3: Comparison: CHA2D2S-VASC Risk Score 1 vs CHA2D2S-VASC Risk Score 4; Test type: Superiority or Other; p = 0.003, Chi-squared; Risk Difference (RD) = 12.4, 95% CI 2-sided [4.7 to 20.1]
Statistical Analysis 4: Comparison: CHA2D2S-VASC Risk Score 1 vs CHA2D2S-VASC Risk Score 5; Test type: Superiority or Other; p = 0.009, Chi-squared; Risk Difference (RD) = 11.1, 95% CI 2-sided [3.2 to 18.8]
Statistical Analysis 5: Comparison: CHA2D2S-VASC Risk Score 1 vs CHA2D2S-VASC Risk Score 2; CHA2D2S-VASC risk score 1 was the reference; Test type: Superiority or Other; p = 0.024, Regression, Logistic; CHA2D2S-VASC risk score 1 was the reference, adjusted for nr diagrams, nr years, age, gender, smb close with stroke, speciality, professional degree; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.08 to 3.07]
Statistical Analysis 6: Comparison: CHA2D2S-VASC Risk Score 1 vs CHA2D2S-VASC Risk Score 3; Test type: Superiority or Other; p = 0.03, Regression, Logistic; Adjusted for age, gender, medical and academic degrees, someone close with stroke, speciality, period of risk estimation, number of figures; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.06 to 2.98] — numerator: CHADS-VASC 1
Statistical Analysis 7: Comparison: CHA2D2S-VASC Risk Score 1 vs CHA2D2S-VASC Risk Score 4; Test type: Superiority or Other; p = 0.002, Regression, Logistic; [statistical method as in outcome 4, analysis 6]; Odds Ratio (OR) = 2.37, 95% CI 2-sided [1.37 to 4.09] — numerator = CHADS-VASC 1
Statistical Analysis 8: Comparison: CHA2D2S-VASC Risk Score 1 vs CHA2D2S-VASC Risk Score 5; Test type: Superiority or Other; p = 0.004, Regression, Logistic; [statistical method as in outcome 4, analysis 6]; Odds Ratio (OR) = 2.19, 95% CI 2-sided [1.14 to 2.56] — numerator=CHADS-VASC 1

ADVERSE EVENTS:
Groups:
- One Diagram: decision aid with one diagram (risk under treatment)
  decision aid: decision aid with one/two diagrams
  OAC prescribed: 400 of 486 (83%)
- Two Diagrams: classical decision aid with 2 diagrams (risk without treatment, and risk with treatment)
  decision aid: decision aid with one/two diagrams
  OAC prescribed: 406 of 482 (83.5%)
Arm/Group | One Diagram | Two Diagrams
Serious Adverse Events (participants affected / at risk) | 0/486 | 0/482
Other Adverse Events (participants affected / at risk) | 0/486 | 0/482

LIMITATIONS AND CAVEATS:
* prescription was only simulated - not real patients, physicians had to imagine they had atrial fibrillation
* results could be different on patients
* participants had to decide prescription/not after seeing the risk diagram for only 5 minutes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No